CLINICAL TRIAL: NCT02418845
Title: A Phase 3, Multi-center, Prospective, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effectiveness and Safety of SYM-1219 2 Grams for the Treatment of Women and Post-Menarchal Adolescent Girls With Bacterial Vaginosis
Brief Title: A Phase 3 Study of SYM-1219 Treatment of Women and Post-Menarchal Adolescent Girls With Bacterial Vaginosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Symbiomix Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYM-1219-301
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYM-1219 (Experimental): Administered orally
  Interventions: Drug: SYM-1219
- Placebo (Placebo Comparator): Administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYM-1219
  Arms: SYM-1219
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to test the safety and efficacy of the oral investigational new drug, SYM-1219 for the treatment of bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Are premenopausal adult females or post menarchal adolescent girls ≥12 years of age in good general health
* Have a clinical diagnosis of bacterial vaginosis, defined as having all of the following criteria:
* Off-white (milky or gray), thin, homogeneous vaginal discharge
* Vaginal pH ≥ 4.7
* Presence of Clue cells of ≥ 20% of the total epithelial cells on microscopic examination of the vaginal saline wet mount
* A positive 10% KOH Whiff test
* Have a Gram stain slide Nugent Score ≥ 4 at the Baseline Visit (Day 1)

Exclusion Criteria:

* Are pregnant, lactating, or planning to become pregnant during the study
* Are menstruating or have vaginal bleeding at the Baseline Visit (Day 1)
* Are suspected clinically (or confirmed diagnostically) of having alternative causes of vaginal symptoms including candidiasis, Chlamydia trachomatis, Trichomonas vaginalis, Neisseria gonorrhoeae or Herpes simplex
* Have received antifungal or antimicrobial therapy (systemic or intravaginal) within 14 days prior to the Baseline Visit (Day 1)

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2015-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Birmingham, Alabama
  - Jonesboro, Arkansas
  - San Diego, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Leesburg, Florida
  - Miami, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Baltimore, Maryland
  - Grand Rapids, Michigan
  - Plainsboro, New Jersey
  - New Bern, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Myrtle Beach, South Carolina
  - Corpus Christi, Texas
  - Houston, Texas
  - Virginia Beach, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female post-menarchal participants age 12 and older, inclusive, with a clinical diagnosis of bacterial vaginosis were recruited and enrolled in 21 investigative medical sites throughout the US. Recruitment/enrollment took place between May 4, 2015 and Sep 24, 2015.
Groups:
- SYM-1219: 2 grams administered orally as a single dose
  SYM-1219
- Placebo: Administered orally as a single dose
  Placebo
Period: Overall Study
Arm/Group | SYM-1219 | Placebo
Started | 125 | 64
Completed | 109 | 52
Not Completed | 16 | 12
Not completed — Lost to Follow-up | 7 | 2
Not completed — Lack of Efficacy | 0 | 3
Not completed — Physician Decision | 5 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Participants deemed eligible at baseline who received a dose from either arm
Groups:
- Total: Total of all reporting groups
Arm/Group | SYM-1219 | Placebo | Total
Number analyzed (Participants) | 125 | 64 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 64 | 189
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 64 | 189
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 12 | 33
  Not Hispanic or Latino | 104 | 52 | 156
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 33 | 100
  White | 55 | 29 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 125 | 64 | 189

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome Responder Rate
Description: Determined by Normal vaginal discharge, negative 10% KOH Whiff test, & Clue cells less than 20%
Time Frame: Study Days 21-30 (End of Study (EOS))
Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who met all inclusion/exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 | Placebo
Number analyzed (Participants) | 107 | 57
Participants
  Clinical Outcome Responder | 57 | 11
  Non-Responder | 50 | 46

2. Secondary Outcome: Clinical Outcome Responder Rate (Interim Visit Only)
Description: Determined by Normal vaginal discharge, negative 10% KOH Whiff test, & Clue cells less than 20%
Time Frame: Study Days 7-14 (interim)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 | Placebo
Number analyzed (Participants) | 107 | 57
Participants
  Clinical Outcome Responder | 62 | 14
  Non-Responder | 45 | 43

3. Secondary Outcome: Gram Stain Slide Nugent Score
Description: A score of 0-3 will be considered normal; a score of 4 and above will be considered abnormal
Time Frame: Study Days 7-14 (interim) & Study Days 21-30 End of Study (EOS)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 | Placebo
Number analyzed (Participants) | 107 | 57
Participants
  Study days 7-14 (interim): Nugent Score 0-3 | 49 | 2
  Study days 7-14 (interim): Nugent Score 4 or greater | 58 | 55
  Study days 21-30 (EOS): Nugent Score 0-3 | 47 | 3
  Study days 21-30 (EOS): Nugent Score 4 or greater | 60 | 54

4. Secondary Outcome: Therapeutic Outcome Responder Rate
Description: A Therapeutic Outcome Responder is defined as a Clinical Outcome Responder with a normal Nugent Score (between 0-3)
Time Frame: Study days 7-14 (interim) & study days 21-30 (EOS)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 | Placebo
Number analyzed (Participants) | 107 | 57
Participants
  Study days 7-14 (interim): Therapeutic Outcome Responder | 37 | 2
  Study days 7-14 (interim): Non-Responder | 70 | 55
  Study days 21-30 (EOS): Therapeutic Outcome Responder | 37 | 2
  Study days 21-30 (EOS): Non-Responder | 70 | 55

5. Secondary Outcome: Investigator's Clinical Assessment
Description: Investigator's opinion of the need for additional Bacterial Vaginosis (BV) treatment (Yes or No)
Time Frame: Study days 21-30 End of Study (EOS)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 | Placebo
Number analyzed (Participants) | 107 | 57
Participants
  Additional BV treatment needed | 32 | 38
  No additional treatment needed | 68 | 16
  Missing | 7 | 3

ADVERSE EVENTS:
Arm/Group | SYM-1219 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/64
Serious Adverse Events (participants affected / at risk) | 2/125 | 0/64
Other Adverse Events (participants affected / at risk) | 43/125 | 14/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYM-1219 (N=125) | Placebo (N=64)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYM-1219 (N=125) | Placebo (N=64)
Vulvovaginal mycotic infection (Infections and infestations) | 9 | 2
Vulvovaginal candidiasis (Infections and infestations) | 8 | 1
Bronchitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Subcutaneous abcess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Nausea (Gastrointestinal disorders) | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 2
Dizziness (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Vulvovaginal pruritis (Reproductive system and breast disorders) | 3 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI submits complete copy of publication material to sponsor at least 60 days prior to submission implementing all reasonable sponsor comments. If sponsor determines that proposed publication contains disclosure of intellectual property for which sponsor is seeking patent protection, PI shall delay submission 60 days from sponsor notice so sponsor may file patent application covering intellectual property. PI shall have no further rights to publish sponsor confidential information.